CLINICAL TRIAL: NCT03422445
Title: A Phase 2 Study of Apatinib Combined With Temozolomide in the Treatment of Advanced Melanoma Patients After Conventional Treatment Failure
Brief Title: A Study of Apatinib Combined With Temozolomide in Patients Witn Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-MEHB002
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Advanced Melanoma
Keywords: Apatinib; Temozolomide; Advanced Melanoma
MeSH Terms: interventions — apatinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus Temozolomide (Experimental): this trial is designed single arm. all the subjects enrolled will receive the experimental intervention,apatinib+temozolomide.
  Interventions: Drug: Apatinib; Drug: Temozolomide

INTERVENTIONS:
Drug: Apatinib — Apatinib：500mg/d，qd，po，d1-28
  Other Names: Apatinib mesylate tablets
Drug: Temozolomide — Temozolomide：300mg/d，qd，po，d1-5

SUMMARY:
30 patients with advanced melanoma will receive apatinib plus Temozolomide as maintenance therapy.

DETAILED DESCRIPTION:
In this study, we plan to enroll 30 patients with advanced melanoma patients who have failed at least one systemic treatment regimen. The therapeutic regimen is temozolomide, 300mg,po, d1-5, apatinib, 500 mg, qd, po, d1-28, Every 28 days for 1 cycles, the primary end point was PFS, the secondary end point was OS, DCR, ORR etc. So we plan to investigate the safety and efficacy of apatinib combined with temozolomide in the treatment of advanced melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old；
* ECOG performance scale 0-1；
* Life expectancy of more than 3 months；
* Histologically or cytologic confirmed melanoma；
* Temozolomide has not been previously treated；
* Patients who have failed at least one systemic treatment regimen： including but not limited to patients receiving immunotherapeutics such as PD-1 monoclonal antibodies, PDL-1 monoclonal antibodies, ipilimumab, C-kit inhibitors, Braf inhibitors, and molecular targeted drugs.
* For results of blood routine test and biochemical tests： Hgb>100g/L, ANC>2.0×109/L, PLT>100×109/L, Serum Total bilirubin ≤ 1.5 X UNL, ALT and AST ≤ 2.5 x upper normal limit (UNL), and ≤ 5 x UNL（Hematogenous metastases）, Serum Creatine ≤ 1.5 x UNL；
* Informed consent；
* Willingness and ability to comply with scheduled visits.

Exclusion Criteria:

* Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)；
* With ≥grade 2 coronary heart disease, arrhythmia (including QTc interval prolongation male ≥450 ms, women ≥470 ms)；
* Imaging studies have shown that the tumor has been infringing on an important perivascular or when the researcher determines that the patient's tumor has a high risk of fatal hemorrhage during treatment；
* Abnormal Coagulation (INR>1.5, PT>UNL+4 seconds), with tendency of bleed or receiving the therapy of thrombolysis or anticoagulation.；
* Urine protein ≥++ or confirmed >1.0 g by the 24h quantity；
* Pregnant and lactating women, or female patients of child-bearing age without taking contraceptive measures；
* A history of psychotropic substance abuse and can not be abstinent or mental disorders ；
* There are serious concomitant diseases that endanger patient safety or affect the patient in completing the study；
* Patients participating in other clinical trials simultaneously；
* Other situations that the researchers considered unsuitable for this study；
* Confirmed brain metastasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival（PFS） | 12 months
  PFS is evaluated in 12 months since the treatment began

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 12 months
  evaluated in the 12th month since the treatment began
Disease Control Rate(DCR) | 12 months
  evaluated in the 12th month since the treatment began
Overall Survival(OS) | 12 months
  evaluated in the 12th month since the treatment began
Safety and Tolerability as measured by adverse events | 12 months
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD，PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou L, Yang Y, Si L, Chi Z, Sheng X, Lian B, Wang X, Tang B, Mao L, Yan X, Li S, Bai X, Guo J, Cui C. Phase II study of apatinib combined with temozolomide in patients with advanced melanoma after failure of immunotherapy. Melanoma Res. 2022 Jun 1;32(3):142-149. doi: 10.1097/CMR.0000000000000809. Epub 2022 Feb 20. PMID 35190519